CLINICAL TRIAL: NCT02679937
Title: Prevention of Obesity in Military Communities - Fit4Duty: Phase 2
Brief Title: Prevention of Obesity in Military Communities - Fit4Duty
Acronym: POMC-Fit4Duty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F172NC-S1
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Overweight; Adiposity
Keywords: U.S. Military; Overweight; Obesity; Service Members; Prevention
MeSH Terms: conditions — Obesity; Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fit4Duty (Experimental): 6-week weight gain prevention group
  Interventions: Behavioral: Fit4Duty
- Nutrition Education (Active Comparator): Two, 50 minute educational videos.
  Interventions: Other: Nutrition Education

INTERVENTIONS:
Behavioral: Fit4Duty — Small (<9) participant-driven groups meet weekly for 6, 1 hour sessions. Participants design small, gradual healthy lifestyle change plans with added verbal, written, and behavioral exercises designed to elicit dissonance regarding engaging in unhealthy eating and sedentary practices. Participants are asked to voluntarily discuss the health, interpersonal and societal costs of obesity, an unhealthy diet, and sedentary behavior, as well as the benefits of leanness, a healthy diet, and regular physical activity.
  Arms: Fit4Duty
Other: Nutrition Education — Two, 50 minute educational videos address basic concepts of healthy nutrition and weight management reviewing topics such as macro and micronutrients, the virtue of whole grains, fruit, vegetables and superfoods, the dangers of dehydration and vitamin deficiency. The role of poor eating habits, lack of exercise and cultural and technological issues in America's obesity epidemic is examined. A basic understanding of energy balance is conveyed. The role of nutritional supplements is addressed.
  Arms: Nutrition Education

SUMMARY:
This randomized controlled trial assesses the efficacy of a 6-week, dissonance-based, weight-gain prevention program (Fit4Duty) designed to reduce unhealthy weight gain among military service members at-risk for obesity. The Fit4Duty program is an adaptation for the military of an existing civilian obesity prevention program, Project Health, which reduced obesity onset by 50% in healthy civilian young adults. Fit4Duty is compared to a nutrition education control condition and is hypothesized to reduce excess weight gain beyond the control comparison program during the 2 year period following study participation.

DETAILED DESCRIPTION:
Obesity is prevalent in military personnel and raises concerns related to health, readiness, and national defense. Adverse health consequences of obesity place military personnel at risk for serious medical problems while in the service and upon discharge/retirement. Additionally, failure to "make weight" may negatively impact one's military career and can lead to discharge from the service. Early identification of personnel at risk and implementation of prevention strategies are critical to addressing the problem of overweight in the military and are essential to maintaining a fit fighting force. The goal of this study is to test the effectiveness of a dissonance-based, weight-gain prevention program (Fit4Duty) to prevent excess weight gain among service members at risk for obesity due to a personal and/or family history of overweight. The Fit4Duty program is an adaptation for the military of an existing civilian obesity prevention program, Project Health. The program utilizes dissonance based, participant-driven group counseling to address the excess consumption of unhealthy foods and sedentary behavior. Active duty service members will be randomized to the Fit4Duty weight gain prevention program or a Nutrition Education comparison condition. Participants will complete height, weight, and body composition measurements, and self-report instruments at baseline, immediately following the prevention program (6-weeks), and one and two year follow-ups. It is hypothesized that Project Fit4Duty will result in significantly greater reduction in risk for increases in BMI percentile and percent fat mass, and risk for onset of overweight and obesity during the 2-year follow-up relative to a nutrition education control program. If successful, Project Fit4Duty would offer an economical approach for widespread obesity prevention in the U.S. Military.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Service Member
* 18.5 kg/m2 < BMI ≤ 32kg/m2
* At risk for excess weight gain due to personal and/or family history of overweight
* English speaking
* Ability to complete study procedures

Exclusion Criteria:

* Presence of a major, chronic medical illness
* Illness and/or treatment likely to affect appetite or body weight
* Planned deployment/ training during the intervention period (upcoming 2 months)
* Documented or self-reported current pregnancy, current breast-feeding, or recently pregnant women (within 1 year of delivery). Because pregnancy is a state in which weight gain is expected and appropriate, pregnant individuals would not be suitable for this study
* Evidence or signs of suicidal ideation as determined by the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12-27 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Participant weight (lbs) | Baseline, Change from basline at post-treatment (6 weeks), 1 year and 2 years
  Participants will be weighed using professional grade equipment and trained personnel

SECONDARY OUTCOMES:
Body Composition: body fat % | Baseline, Change from basline at post-treatment (6 weeks), 1 year and 2 years
  Participants' body composition will be determined using professional grade equipment and trained personnel
Abdominal waist and hip circumference | Baseline, Change from basline at post-treatment (6 weeks), 1 year and 2 years
  Participants will be measured using a cloth tape measure with a spring-loaded handle

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Sbrocco, PhD, Principal Investigator — Uniformed Services University of the Health Sciences; Douglas Maurer, DO, MPH, Principal Investigator — Madigan Army Medical Center
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No